CLINICAL TRIAL: NCT06332040
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Gentamicin Bladder Instillation on CAUTI
Brief Title: Gentamicin Bladder Instillation on CAUTI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-500-243-50-35
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Catheter Infection
MeSH Terms: interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gentamicin (Experimental): 14.4 mg gentamicin dissolved in 30 mL 0f 0.9% saline administered BID
  Interventions: Drug: Gentamicin
- Placebo (Placebo Comparator): 30 mL of 0.9% saline administered BID
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Gentamicin — random assignment to gentamicin or placebo bladder instillation to prevent CAUTI (catheterized urinary track infection)

SUMMARY:
Urinary tract infections in catheterized patients is an unacceptable complication and has been termed a 'never event' by the Center for Medicare & Medicaid Services (CMS); however there is not consensus among clinicians on how to best prevent CAUTIs. We propose a prospective randomized controlled trial to test the efficacy of prophylactic gentamicin bladder irrigation in elimination of CAUTIs.

DETAILED DESCRIPTION:
Catheter Associated Urinary Tract Infection (CAUTI) is a hospital acquired infection considered preventable by the Center for Medicare & Medicaid Services (CMS) and originally estimated to cost each individual patient approximately $4700 per infection in 2009 US dollars1. In the inpatient population, more contemporary calculations have associated the per patient cost to have risen to a mean of $13,793 per patient (range $4,694-$29,743)2, with an increased median length of stay of 3.6 days, and a 1.37 increased odds ratio of death3.

CMS understandably has declared CAUTI a "never event", a term coined by the National Quality Forum and used to describe preventable hospital acquired infections4. Since 2008 they have tied this quality metric to severe hospital payment penalties to incentivize prioritization of strategies to decrease CAUTIs.

Despite considerable efforts to remain in compliance with this guidance, and hospitals nationwide implementing safer catheter placement training as well as aggressive early catheter removal protocols, it has become clear that CAUTIs are almost never a never event5. Quantitative analyses of these events have estimated that only 65-70% of CAUTIs are truly preventable with current evidence-based prevention strategies6.

In our intensive care units the pragmatic reasons explaining this phenomenon are abundantly clear. Trauma patients critically injured with multiple spinal, pelvic and long bone fractures, intubated on a ventilator and immobile have substantially higher rates of urine retention when foley catheters are removed aggressively within 72 hours of admission per current infection control protocols. Similarly, neuro critical care patients who incurred a massive stroke or traumatic brain injury who are immobilized from their disabilities do not routinely succeed with early catheter removal protocols. Replacing indwelling foley catheters after multiple failed intermittent urinary catheterizations incurs increased urethral trauma and pain for the patient, increased risk of procedural complications, and increased risk of CAUTI due to repeated urethral instrumentation.

On the basis of and in response to a clear need to develop novel strategies to eliminate CAUTIs in those patients for whom early catheter removal is not deemed clinically appropriate, we collected 8 months of pilot data at our level I trauma center ICU in which we prophylactically instilled an antibiotic containing irrigation solution into the indwelling foley catheters in patients who required catheterization for greater than 3 days. Over the observed pilot period zero CAUTI events were recorded as compared to a comparison control group of trauma patients with identical inclusion criteria for whom 9 "never event" CAUTIs were incurred. These differences were statistically significant.

The current proposal aims to expand this pilot data and conduct a full randomized trial to validate the efficacy of gentamicin antibiotic irrigation in critically ill patients with an indwelling foley catheter of greater than 3 days duration. We plan to expand our patient population to include critically ill patients admitted to the trauma, neuro-critical care and medical ICU units.

The current proposal aims to expand this pilot data and conduct a randomized trial to validate the efficacy of gentamicin antibiotic irrigation in critically ill patients with an indwelling foley catheter of greater than 3 days duration. We plan to expand our patient population to include critically ill patients admitted to the trauma, neuro-critical care and medical ICU units. Our primary research question is: Is prophylactic gentamicin bladder irrigation associated with decreased CAUTI in a cohort of catheterized trauma and neuro critical care patients.

ELIGIBILITY:
Inclusion Criteria:

1. age greater than 18
2. admitted with a trauma, surgical, or neuro-critical care diagnosis
3. indwelling foley catheter in place

Exclusion Criteria:

1. Documented positive UA or Urine Culture within the past 7 days or upon admission
2. Traumatic bladder injury
3. Gross hematuria
4. Chronic indwelling urethral or chronic suprapubic foley catheter
5. allergy to gentamicin or similar aminoglycosides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
CAUTI as primary outcome | 30 days
  positive urine culture

CONTACTS AND LOCATIONS:
Overall Officials: Hahn Soe-Lin, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix
Locations (1):
- St. Jpseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No